CLINICAL TRIAL: NCT04238312
Title: The Effect of a Respiratory Biofeedback Device on Reduction of Dental Anxiety Associated With Local Anesthesia in Children: A Randomized Controlled Clinical Trial
Brief Title: Respiratory Biofeedback Device and Reduction of Dental Anxiety Associated With Local Anesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health and Statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Respiratory biofeedback device
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study will be a randomized controlled clinical trial, with 1:1 allocation ratio.
Masking Description: The operator will not be blinded to the treatment as the RESPeRATE™ will be used for the study group while the device will not be applied to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESPeRATE™ (Experimental): RESPeRATE™: 2breathe Tech. Ltd., Eshtaol, Israel. The device includes a belt-type respiration sensor worn outside of the clothing that is placed around the torso. It is connected to a computerized box that generates musical patterns listened through an earbud. The device guides the user interactively to slow breathing with a relatively prolonged expiration.
  Interventions: Device: RESPeRATE™
- Tell, Show and Do technique (Active Comparator)
  Interventions: Behavioral: Tell, Show and Do technique

INTERVENTIONS:
Device: RESPeRATE™ — Fifty-five anxious pediatric dental patients received a breathing session of 10 minutes, using the RESPeRATE™ device.
  Arms: RESPeRATE™
Behavioral: Tell, Show and Do technique — Fifty-five anxious pediatric dental patients received a traditional behavior management technique (Tell-Show-Do).
  Arms: Tell, Show and Do technique

SUMMARY:
The aim of the study was to investigate the effect of a respiratory biofeedback device (RESPeRATE TM) in reduction of preoperative anxiety in children undergoing dental procedures under local anesthesia.

DETAILED DESCRIPTION:
The study was a randomized controlled clinical trial. A total of 110 anxious pediatric dental patients, of age range 7-12 years, were selected from the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, Egypt, after securing parental informed consents. Children were chosen according to the Faces version of Modified Child Dental Anxiety Scale scoring 26 or more.

The participants will be randomly allocated into 2 groups: Group I: Study group and Group II: Control group. The patients of group I (Study group) will undergo a session of biofeedback regulation by using "RESPeRATETM" as an anxiety reducing method. Group II patients will be managed by a routine behavioral management technique "Tell,show,do". Local anesthesia injection will be administered to the child, after which heart rate measurement and salivary sample for salivary amylase analysis will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy children (physical status ASA I & II).
* Scoring 26 or more on faces version of modified child dental anxiety scale (MCDASf).
* Dental procedure requiring local anesthesia.
* Completion of a parental consent to participate in the study.

Exclusion Criteria:

* Children on anxiolytic medication or using any medication directly related to emotional or cognitive function.
* Children with special needs.
* Children on medications that specifically agonize or antagonize alpha- or beta-adrenergic processes.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Heart Rate | baseline
  A finger pulse oximeter will be placed on the finger of the left hand of the child.
Heart Rate | after 5 minutes
  A finger pulse oximeter will be placed on the finger of the left hand of the child.
Oxygen saturation | baseline
  Oxygen saturation will be monitored using an oximeter
Oxygen saturation | after 5 minutes
  Oxygen saturation will be monitored using an oximeter
Behavior Evaluation | baseline
  using Frankl scale (ranges from 1-4); 1: Definitely negative, 2: negative, 3:positive and 4: definitely positive
Behavior Evaluation | after 1 week during follow-up sessions
  using Frankl scale (ranges from 1-4); 1: Definitely negative, 2: negative, 3:positive and 4: definitely positive

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Zeitoun, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Amani Khalil, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Nadia Wahba, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Mohamed IS Ahmed, PhD, Study Chair — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Morarend QA, Spector ML, Dawson DV, Clark SH, Holmes DC. The use of a respiratory rate biofeedback device to reduce dental anxiety: an exploratory investigation. Appl Psychophysiol Biofeedback. 2011 Jun;36(2):63-70. doi: 10.1007/s10484-011-9148-z. PMID 21365307
- [Background] Howard KE, Freeman R. Reliability and validity of a faces version of the Modified Child Dental Anxiety Scale. Int J Paediatr Dent. 2007 Jul;17(4):281-8. doi: 10.1111/j.1365-263X.2007.00830.x. PMID 17559456
- [Background] Chipps J. Psychological therapies for the management of chronic and recurrent pain in children and adolescents: A Cochrane review summary. Int J Nurs Stud. 2021 Jan;113:103393. doi: 10.1016/j.ijnurstu.2019.103393. Epub 2019 Aug 16. No abstract available. PMID 31519334